CLINICAL TRIAL: NCT05895357
Title: The Effect of Music Therapy on Comfort, Pain and Anxiety in Patients With Bone Marrow Aspiration and Biopsy: A Randomized Controlled Research
Brief Title: The Effect of Music Therapy on Comfort, Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, seda şahan, Phd research assistant, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 820
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Bone Marrow Disease; Hematological Malignancy
Keywords: bone marrow; aspiration; biopsy; musictherapy; anxiety; pain; comfort
MeSH Terms: conditions — Bone Marrow Diseases; Hematologic Neoplasms; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): The patients were asked about the type of music they wanted to listen to. Especially in the last meta-analyses, it was determined that listening to the music that patients chose was more effective (Witten 2020). For this reason, after the intervention group is asked about the music they want to listen to, the music they want will be played from the music application.
  Interventions: Other: Musictherapy
- No intervention (No Intervention): The patients in the control group will not listen to music, and routine procedures will performed in the clinic without additional intervention. Anxiety, pain, and comfort assessments will made in the control group patients before and after the procedure.

INTERVENTIONS:
Other: Musictherapy — The patients were asked about the type of music they wanted to listen to. Especially in the last meta-analyses, it was determined that listening to the music that patients chose was more effective (Witten 2020). For this reason, after the intervention group is asked about the music they want to listen to, the music they want will be played from the music application.
  Arms: Music Therapy

SUMMARY:
Objectives: This study was conducted to determine the effect of music therapy on the pain, anxiety, and comfort levels of patients who underwent bone marrow aspiration and biopsy.

Methods: This research was conducted as a randomized controlled study in the hematology polyclinic of a university hospital. Music therapy will used with the intervention group throughout the procedure. During data evaluation, paired t-test, independent t-test and effect size will used. The sample group was calculated based on the sample groups of other studies in the literature (Çelebi et al., 2020; Özdemir et al., 2019). According to the preliminary power analysis results using the G.Power 3.1.9 program, the sample size was calculated at 80% power, at medium effect size at 5% alpha value. According to the analysis results, the sample size per group was calculated as 30. However, since there was 10% probability that some patients may drop, the sample size for the study was recalculated as 66 (Experimental Group: 33, Control Group: 33).The patients will informed about using music. In addition, it will explained that they could adjust the sound levels and that they should report when they are disturbed by the tone. Music continued throughout the process. Communication with the patient will maintained, and symptoms such as discomfort, anxiety were observed throughout the procedure. The music player will switched off after the procedure was completed. The patients will asked whether they had any discomfort while the music played. TThe music therapy will last an average of 30 minutes. After completing the procedures, the patient's pain, comfort, and anxiety levels were re-evaluated using VAS and STAI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hematological malignancy (defined as multiple myeloma, Chronic Lymphocytic Leukaemia, Myelodysplastic syndrome or indolent lymphoma)
* 18 years of age or older,
* Must be able to speak Turkish

Exclusion Criteria:

* Hearing impairment
* hormonal dysfunction (adrenal, pituitary, thyroid, etc.)
* Sever anxiety disorder
* Parkinson's disease
* Alzheimer's disease
* Dementia
* Major depression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain and Comfort | 10 minutes
  The scale, used to measure patients' subjective pain and comfort, was developed by Price et al. (1983) (Price et al., 1983). This scale consists of a 10 cm horizontal or vertical line with both ends representing the minimum and maximum scores for pain and comfort (0: no pain/no discomfort (very comfortable), 10: most severe pain/very uncomfortable (not at all). Comfort was defined by patients as a pleasant feeling and as the absence of physical discomfort. The patients will asked to indicate their pain severity and comfort on the scale. The distance between the indicated point and the lowest endpoint of the line will measured in centimeters using a ruler, and the numeric value will assigned as the individual's pain score.

SECONDARY OUTCOMES:
State Trait Anxiety Scale (STAI) | 10 minutes
  The inventory consisting 40 items was developed by Spielberger et al. (1983) (Spielberger, 1983). The STAI consists of two separate scales to assess state (STAI-S) and trait (STAI-T) anxiety. Öner (1998) performed the Turkish validity and reliability studies of the scale. In the validity and reliability study of the STAI Turkish form, test-retest reliability coefficients ranged from 0,94 to 0,96 for state anxiety and ranged from 0,83 and 0,87 for trait anxiety. The State Anxiety Inventory with 20 items (Items 1-20) that assess the respondent's current feelings was used in this study. Each item is rated on a 4-point Likert scale from 1 (Almost never) to 4 (Almost always). Subscale scores range from 20 to 80, and higher scores indicate higher anxiety levels

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Other researchers can get information by sending an e-mail to the responsible researcher of this study. (seda.sahan@bakircay.edu.tr)

REFERENCES:
- [Derived] Sahan S, Korkmaz E, Korkmaz S. The effect of music on comfort, pain, and anxiety in patients with bone marrow aspiration and biopsy in Turkey: a mixed-methods study. BMC Complement Med Ther. 2024 Jun 12;24(1):228. doi: 10.1186/s12906-024-04531-0. PMID 38867235